CLINICAL TRIAL: NCT00545779
Title: 'Open, Prospective, Multi-center, Two-part Study of Patient Preference With Monthly Ibandronate Therapy in Women With Postmenopausal Osteoporosis Switched From Once-daily or Once Weekly Alendronate or Risendronate - BONCURE (BONviva for Current Bisphosphonate Users - Regional European Trial)'
Brief Title: BONCURE Study: A Study of Monthly Bonviva (Ibandronate) in Women With Post-Menopausal Osteoporosis on Bisphosphonate Therapy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20430
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Results first posted 2016-10-28 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-09

CONDITIONS: Post-Menopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Ibandronic Acid

ARMS (1):
- Ibandronate (Experimental): Participants completed Candidate Identification Questionnaire (CIQ) in Part A and received Ibandronate 150 milligram (mg) tablet orally once-monthly up to 6 months in Part B of the study.
  Interventions: Drug: Ibandronate

INTERVENTIONS:
Drug: Ibandronate — 150 mg orally once monthly for 6 months
  Other Names: [Bonviva/Boniva]

SUMMARY:
This single arm study will assess participant preference for monthly Bonviva, versus daily or weekly alendronate or risedronate, in the treatment of postmenopausal osteoporosis. Participants currently on a daily or weekly regimen of bisphosphonate therapy (alendronate or risedronate) will answer a questionnaire to identify participants who may benefit from a monthly Bonviva regimen. Eligible participants will then discontinue their present bisphosphonate treatment, and switch to monthly Bonviva 150mg per oral (po). At the beginning and end of Bonviva treatment, all participants will complete an Osteoporosis Patient Satisfaction Questionnaire. The anticipated time on study treatment is 3-12 months, and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* post-menopausal women;
* >=3 months daily or weekly alendronate or risedronate for treatment or prevention of post-menopausal osteoporosis.

Exclusion Criteria:

* inability to stand or sit in an upright position for at least 60 minutes;
* hypersensitivity to bisphosphonates;
* treatment with other drugs affecting bone metabolism;
* abnormalities of the oesophagus, which delay oesophageal emptying.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 677 (Actual)
Dates: Start 2006-12; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (27):
- Tirana, Albania
- Bosnia and Herzegovina (3):
  - Banja Luka
  - Sarajevo
  - Tuzla
- Croatia (4):
  - Rijeka
  - Slavonski Brod
  - Split
  - Zagreb
- Skopje, North Macedonia
- Serbia (3):
  - Belgrade
  - Niška Banja
  - Novi Sad
- Turkey (Türkiye) (15):
  - Adana
  - Ankara
  - Antalya
  - Aydin
  - Bursa
  - Denizli
  - Erzurum
  - Gaziantep
  - Istanbul
  - Izmir
  - Kayseri
  - Konya
  - Manisa
  - Samsun
  - Trabzon

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ibandronate
Started | 677
Completed | 633
Not Completed | 44
Not completed — Violation of selection criteria at entry | 8
Not completed — Other protocol violation | 1
Not completed — Did not cooperate | 7
Not completed — Withdrawal by Subject | 20
Not completed — Adverse Event/intercurrent illness | 5
Not completed — Failure to return | 3

BASELINE CHARACTERISTICS:
Population: Analysis population included all enrolled participants in Part A who provided the baseline information.
Arm/Group | Ibandronate
Number analyzed (Participants) | 670
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 670
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Current Daily or Weekly Bisphosphonate Users in Part A Who Answer 'Yes' to Any of the Questions in the Candidate Identification Questionnaire (CIQ)
Description: The CIQ was completed in Part A by all the participants. The information from the CIQ was used to determine the percentage of current daily or weekly bisphosphonate users for whom monthly ibandronate represented a potentially more satisfactory therapeutic option.
  In the CIQ participants were asked to answer either 'yes' or 'no' to the following 3 questions:
  1. I would prefer a monthly oral dosing schedule to my current (daily or weekly) dosing schedule.
  2. More than once per month, I have experienced stomach upset within 48 hours of taking my osteoporosis medication.
  3. Over the past 3 months, I have missed taking 3 or more doses of my current (daily or weekly) osteoporosis medication.
Time Frame: Visit 0 (less than or equal to [<=] Day -30)
Population: All enrolled participants who completed the part A of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Ibandronate
Number analyzed (Participants) | 677
percentage of participants | 68.1

2. Primary Outcome: Percentage of Participants Who Reported Preference for Monthly Ibandronate
Description: Percentage of participants who reported preference for monthly ibandronate were reported.
Time Frame: Visit 0 (<= Day -30)
Population: All enrolled participants who completed the part A of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Ibandronate
Number analyzed (Participants) | 677
percentage of participants | 67.5

3. Primary Outcome: Percentage of Participants With Positive Change in Total Composite Satisfaction Score (CSS) at Month 6 in Part B by CIQ Fracture (Fr) Group
Description: Participants with a positive change from their baseline CSS at Month 6 are considered those participants who are satisfied with once-monthly dosing of ibandronate after 6 months of use were reported. The CSS is scaled from 0 to 100 and is an average of the 4 domain scores of the Osteoporosis Patient Satisfaction Questionnaire (OPSAT-Q): Convenience (questions 1 to 6), Quality of Life (questions 7 and 8), Overall Satisfaction (questions 9 and 10) and Side Effects (questions 11 to 16). Higher scores indicating greater satisfaction.
Time Frame: Month 6
Population: The intent-to treat (ITT) population included all participants who received at least one dose of study medication. Number of participant analyzed are with or without previous history of Fr.
Measure: Number; unit: percentage of participants
Arm/Group | Ibandronate
Number analyzed (Participants) | 627
percentage of participants
  Participants answer Yes with previous Fr (n=115) | 86.1
  Participants answer Yes without previous Fr(n=310) | 89.0
  Participants answer NO with previous Fr (n=47) | 87.2
  Participants answer NO without previous Fr (n=155) | 77.4

4. Secondary Outcome: Percentage of Participants Eligible Current Daily or Weekly Bisphosphonate Users at Screening Who Elect to Enter Part B by CIQ
Time Frame: Visit 0 (<= Day -30)
Population: The ITT population included all participants who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Ibandronate
Number analyzed (Participants) | 645
percentage of participants
  Answered Yes to at least 1 question in CIQ | 68.1
  Answered NO to every question in CIQ | 31.9

5. Secondary Outcome: Percentage of Participants Who Reported an Improved Satisfaction Score After 6 Months in Part B
Description: Percentage of participants who report an improved satisfaction score after 6 months of monthly ibandronate therapy as compared to daily or weekly alendronate or risendronate at baseline based on responses to each individual question in the CIQ were reported. In the CIQ participants were asked to answer either 'yes' or 'no' to the following 3 questions:
  1. I would prefer a monthly oral dosing schedule to my current (daily or weekly) dosing schedule
  2. More than once per month, I have experienced stomach upset within 48 hours of taking my osteoporosis medication
  3. Over the past 3 months, I have missed taking 3 or more doses of my current (daily or weekly) osteoporosis medication
Time Frame: Month 6
Population: The ITT population included all participants who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Ibandronate
Number analyzed (Participants) | 645
percentage of participants
  CIQ Question 1 = Yes (n=422) | 88.2
  CIQ Question 1 = No (n=205) | 80.0
  CIQ Question 2 = Yes (n=115) | 93.0
  CIQ Question 2 = No (n=512) | 83.8
  CIQ Question 3 = Yes (n=97) | 94.8
  CIQ Question 3 = No (n=530) | 83.8

6. Secondary Outcome: Percentage of Participants Who Have Greater Than or Equal to (>=) 80% Compliance With 6 Monthly Doses of Ibandronate in Part B
Time Frame: Up to Month 6
Population: The ITT population included all participants who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Ibandronate
Number analyzed (Participants) | 645
percentage of participants | 98.6

7. Secondary Outcome: Percentage of Participants Who Choose a Monthly Reminder to Take Ibandronate in Part B
Time Frame: Visit 0 (<= Day -30)
Population: The ITT population included all participants who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Ibandronate
Number analyzed (Participants) | 645
percentage of participants | 99.4

8. Secondary Outcome: Percentage of Participants Who Reported an Improvement in the Frequency of Gastro-intestinal (GI) Symptoms Per Month in Part B
Time Frame: Baseline to Month 6
Population: Analysis was not performed because the data were difficult or impossible to derive from the database.
Arm/Group | Ibandronate
Number analyzed (Participants) | 0

9. Secondary Outcome: Percentage of Participants by Age and Activity Level Reporting High Satisfaction According to the Osteoporosis Patient Satisfaction Questionnaire (OPSAT-Q) in Part B
Time Frame: Month 6
Population: Analysis was not performed because the data were difficult or impossible to derive from the database.
Arm/Group | Ibandronate
Number analyzed (Participants) | 0

10. Secondary Outcome: Osteoporosis Patient Satisfaction Questionnaire (OPSAT-Q) Domain Scores in Part B
Description: The OPSAT-Q is a validated questionnaire designed to capture satisfaction with bisphosphonate treatment. It comprises four domains: convenience (questions 1-6), quality of life (questions 7 and 8), overall satisfaction (questions 9 and 10), and side effects (questions 11-16). Each domain (scale) ranges 0-100 scale. All items were scored such that higher scores represented greater satisfaction or less bother. Treatment satisfaction was measured with the OPSAT-Q composite satisfaction score (OPSAT-Q CSS), which was the average of the scores from the four domains of the OPSAT-Q converted to a 0-100-point scale, in which higher scores indicate greater satisfaction.
Time Frame: Baseline, Month 6
Population: The ITT population included all participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ibandronate
Number analyzed (Participants) | 645
units on a scale
  Baseline: Convenience | 58.4 (25.4)
  Month 6: Convenience | 89.2 (11.2)
  Baseline: Confidence with daily functioning | 62.6 (25.6)
  Month 6: Confidence with daily functioning | 86.6 (14.8)
  Baseline: Overall satisfaction | 61.4 (27.0)
  Month 6: Overall satisfaction | 89.1 (14.9)
  Baseline: Side effects | 83.7 (91.7)
  Month 6: Side effects | 93.2 (14.2)

ADVERSE EVENTS:
Time Frame: Baseline (Visit 1 of Part B) up to 15 days after the final visit (Month 6)
Description: The Safety Population included 640 participants, who continued into Part B of the study and took at least one dose of study medication.
Arm/Group | Ibandronate
Serious Adverse Events (participants affected / at risk) | 6/640
Other Adverse Events (participants affected / at risk) | 18/640
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibandronate (N=640)
Pericarditis (Cardiac disorders) | 1
Iridocyclitis (Eye disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Hiatus hernia (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Postoperative hernia (Injury, poisoning and procedural complications) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ibandronate (N=640)
Dyspepsia (Gastrointestinal disorders) | 12
Nausea (Gastrointestinal disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.